CLINICAL TRIAL: NCT02613416
Title: Phase II Correlative Study of Denosumab Effects on Tissue and Imaging Breast Biomarkers
Brief Title: Denosumab and MRI Breast Imaging
Acronym: Dmab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alison Stopeck (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, Alison Stopeck, Professor of Medicine, Stony Brook University
Organization: Stony Brook University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 706513
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Denosumab (Experimental): 6 monthly subcutaneous injections of denosumab
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab — monthly subcutaneous injections
  Other Names: XGEVA

SUMMARY:
This is a non-randomized phase II trial of denosumab at 120 mg subcutaneous injection monthly in pre- and post-menopausal women diagnosed with stage 0-III breast cancer who are currently not receiving anticancer treatment with hormonal therapies, chemotherapy, or radiation. All patients will undergo quantification of breast density by MRI at baseline and after 6 months on denosumab. Because the therapeutic agent is an injectable drug, the investigators will conduct a single arm study with both pre- and post-treatment measurements to determine the extent of variability in breast density over time and a placebo treatment period or group will not be utilized. This is an investigator initiated trial and Amgen (SPONSOR) will provide the trial drug denosumab.

DETAILED DESCRIPTION:
According to the results of several studies footnoted in this protocol, there is now convincing evidence that extensive areas of radiographically-dense tissue in the breast is an independent risk factor for the development of breast cancer. Here, the investigators postulate that it is RANK ligand that mediates the association between breast density and risk of breast cancer for which progesterone is one of several factors that influence the availability of RANK ligand in mammary tissue to promote or sustain higher breast density. As such, the investigators hypothesize that inhibition of RANK ligand with the anti-RANK ligand antibody therapeutic agent denosumab will decrease breast density; a risk factor for breast cancer development. The investigators will test the primary hypothesis that RANK ligand inhibition by denosumab (Xgeva) given 120mg monthly to pre- and post-menopausal breast cancer patients will significantly decrease breast density over 6 months. Breast density will be assessed by magnetic resonance fat water imaging (MR-FW) of the breast. At the beginning of the study participants will be measured for a change in breast density by MRI between baseline 1 and baseline 2 (end of 3 months observation period). All patients will then receive 6 months of 120 mg denosumab subcutaneously every month with repeat MR imaging to obtain measurements after 6 months on denosumab. All participants will be asked to provide an optional core needle breast biopsy sample at baseline and after 6 months on denosumab.

ELIGIBILITY:
Inclusion Criteria:

* Pre or postmenopausal women with first incidence of early stage (stages 0 - III) breast cancer who have completed all treatment and are cancer-free, which includes women at high risk for developing invasive cancer i.e. having a breast biopsy positive for atypical ductal or lobular hyperplasia or carcinoma in situ.
* Age ≤ 75 years
* 44 patients will be accrued as follows: a) 22 evaluable patients will be premenopausal as defined as regular menses (24-38 days) b) 22 evaluable patients will be postmenopausal as defined by a history of amenorrhea for at least one year or hormone levels (estradiol/FSH) consistent with menopause if post-hysterectomy status, or history of surgical/medical castration.
* Normal serum calcium or albumin-adjusted serum calcium between 2.0 and 2.9 mmol/L (8.0-11.5mg/dL).
* Adequate vitamin D level (25-hydroxy vitamin D level > 20 ng/mL)
* Currently on no active treatment for breast cancer and at least 3 months post all the treatments, with the exception of aromatase inhibitors (exemestane, anastrozole, letrozole)
* No prior or current use of IV bisphosphonates
* No current use of oral bisphosphonates
* Patients must have an unaffected, non-irradiated contralateral breast
* Significant breast density as determined by mammography and defined by the descriptive terms scattered fibroglandular tissue/densities, heterogeneously dense, or mostly dense tissue in the mammography report.
* Adequate renal function defined as a serum creatinine < 1.5 x ULN or CrCl > 30mL/min
* A willingness and ability to follow the study protocol, as indicated by provision of informed consent to participate
* Willingness to being tested for current pregnancy and use of birth control while being treated with denosumab (pre-menopausal women only)

Exclusion Criteria:

* Age > 75 years
* Subject has known sensitivity to any of the products to be administered during the study (e.g., mammalian derived products, denosumab, calcium, or vitamin D).
* Patients have prior history or current evidence of osteonecrosis or osteomyelitis of the jaw.
* Patients have active dental or jaw condition which requires oral surgery, including tooth extraction.
* Patients have non-healed dental or oral surgery, including tooth extraction.
* Patients with planned invasive dental procedures
* Subject is pregnant or breast feeding, or planning to become pregnant within 5 months after the end of the treatment
* Subject is of child bearing potential and is not willing to use, in combination with her partner, highly effective methods of contraception or abstinence during treatment and for 5 months after the end of treatment
* Active infection with Hepatitis B, Hepatitis C, or Human Immunodeficiency virus (HIV)
* Any condition or disorder that compromises the ability of the subject to provide written informed consent and/or comply with study procedures
* History of claustrophobia
* Have electrically, magnetically, or mechanically activated implants including cardiac pacemaker, cochlear implants, magnetic surgical clips or prostheses.

Max Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-11; Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Stopeck, MD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University Cancer Center, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 12 consented patients were determined to be eligible but withdrew consent before the start of the study intervention
Groups:
- Denosumab 120 mg Subcutaneous: 6 monthly subcutaneous injections of denosumab
  Denosumab: monthly subcutaneous injections
Period: Overall Study
Arm/Group | Denosumab 120 mg Subcutaneous
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Denosumab
Number analyzed (Participants) | 30
Age, Continuous [Median (Standard Deviation); unit: years] | 59.5 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30
Percentage of Breast Density by Magnetic Resonance Imaging [Median (Full Range); unit: percent] | 19.74 [7.85 to 48.62]

OUTCOME MEASURES:

1. Primary Outcome: Relative Change of ≥ 5% in Breast Density at 6 Months
Description: Breast density will be measured via non-contrast MRI before and after 6 months on denosumab
Time Frame: baseline, 6 months
Population: 5 subjects were excluded (ineligible (n=1), withdrew consent (n=1), implants both breasts (n=1) and image artifacts (n=2).
Measure: Count of Participants; unit: Participants
Arm/Group | Denosumab 120 mg Subcutaneous
Number analyzed (Participants) | 25
Participants
  Decrease in breast density of ≥ 5% at 6 months | 13
  No change in breast density | 8
  Increase in breast density of ≥ 5% at 6 months density | 4
Statistical Analysis 1: Comparison: Denosumab 120 mg Subcutaneous; The primary hypothesis for this early phase study was that at least 30% of women would experience a >5% relative decrease in their breast density after 6 months of treatment with denosumab 120 mg subcutaneous dose once a month; Test type: Other; p = 0.026, Blyth-Still Casella Confidence Interval — The p value was calculated

2. Secondary Outcome: Absolute Change > 1% in Breast Density
Description: Unadjusted Absolute Change > 1% in breast density
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Denosumab 120 mg Subcutaneous
Number analyzed (Participants) | 25
Participants
  >1% decrease in breast density | 13
  no change in breast density | 8
  >1% increase in breast density | 4

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Denosumab
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT02613416/Prot_SAP_000.pdf